CLINICAL TRIAL: NCT02432248
Title: Effect of Dehydroepiandrosterone on Live Birth Rate in Subfertile Patients With Poor Ovarian Responds
Brief Title: Effect of DHEA on Patients With Poor Ovarian Responds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S00056W9
Record Dates: First submitted 2015-03-17; First posted 2015-05-04 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Subfertility
Keywords: DHEA; live birth rate; poor ovarian responder
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dehydroepiandrosterone (Experimental): DHEA is considered as health supplement and is available over the counter. Side effects are minimal at present dosage (25mg or 50mg tds).
  Interventions: Drug: Dehydroepiandrosterone
- Placebo (Placebo Comparator): Medical starch is considered as medicine components. Side effects are minimal at present dosage.
  Interventions: Other: placebo(medical starch)

INTERVENTIONS:
Drug: Dehydroepiandrosterone — 75mg/day, PO for 90 days
  Other Names: DHEA
  Arms: Dehydroepiandrosterone
Other: placebo(medical starch) — 75mg/day, PO for 90 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of DHEA for treatment of subfertile patients with poor ovarian reserve and post-treatment evaluation of IVF outcome.

DETAILED DESCRIPTION:
The aim of this randomized controlled study is to compare the effect of DHEA and placebo on live birth rate in poor ovarian responders. Consecutive infertile women attending the subfertility clinic for IVF treatment will be approached. Those fulfilling the selection criteria would be recruited and a written consent will be obtained after detailed explanation and counseling.

Baseline assessment will be performed at early follicular phase (Day 2 or 3) at recruitment. Patient characteristics including age, body mass index (BMI), and smoking status would be recorded and blood test including follicular stimulating hormone (FSH), estradiol (E2), testosterone and anti-Müllerian hormone (AMH) would be checked. Pelvic scan will be performed to assess the total antral follicle count (AFC) and total ovarian volume.

Subjects will be randomized divided into two groups:

1. DHEA group: Subjects will take DHEA (Vitacost) 25mg three times a day for 12 weeks prior to the start of IVF treatment.
2. Placebo group: Subjects will take placebo three times a day for 12 weeks prior to the start of IVF treatment.

Ultrasound assessment will be repeated in follicular phase (D2 or 3) of every month or cycle followed by a IVF treatment using antagonist protocol based on our standard departmental regimen. Cycle characteristics including the dose of gonadotrophins use, duration of stimulation, number of oocytes obtained, number of fertilized embryos and good quality embryos will be recorded and follicular fluid will be saved for hormonal profiles.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for IVF treatment according to our standard department protocol
* Age < 42
* Regular menstrual cycles (21-35 days)

Poor ovarian responders are defined according to the Bologna criteria fulfilling 2 out of 3 of the following:

* Advanced maternal age (≥40) or any other genetic or acquired risk factor for POR
* Previous poor ovarian response (POR) (≤3 oocytes with a conventional stimulation protocol using at least 150IU gonadotrophins per day)
* Abnormal ovarian reserve test (i.e. AFC < 5-7 or AMH < 0.5-1.1ng/ml). Alternatively, two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ORT.

Exclusion Criteria:

* Previous chemotherapy or pelvic irradiation
* Polycystic ovarian syndrome or polycystic ovaries
* On hormonal supplementation for any indication at the time of recruitment (e.g. estrogen, testosterone or DHEA)

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-02; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Participants will be followed for live birth rate up to 1 year.
  Compare the live birth rate between DHEA group and placebo group

SECONDARY OUTCOMES:
Pregnancy rate | Participants will be followed for pregnancy rate up to 1 year.
  Compare the pregnancy rate between DHEA group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, PHD, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University
Locations (1):
- The Affiliated Hospital of Inner Mongolia Medical University, Inner Mongolia, China

REFERENCES:
- [Background] Ubaldi FM, Rienzi L, Ferrero S, Baroni E, Sapienza F, Cobellis L, Greco E. Management of poor responders in IVF. Reprod Biomed Online. 2005 Feb;10(2):235-46. doi: 10.1016/s1472-6483(10)60946-7. PMID 15823231
- [Background] Arlt W, Justl HG, Callies F, Reincke M, Hubler D, Oettel M, Ernst M, Schulte HM, Allolio B. Oral dehydroepiandrosterone for adrenal androgen replacement: pharmacokinetics and peripheral conversion to androgens and estrogens in young healthy females after dexamethasone suppression. J Clin Endocrinol Metab. 1998 Jun;83(6):1928-34. doi: 10.1210/jcem.83.6.4850. PMID 9626121
- [Background] Shifren JL, Braunstein GD, Simon JA, Casson PR, Buster JE, Redmond GP, Burki RE, Ginsburg ES, Rosen RC, Leiblum SR, Caramelli KE, Mazer NA. Transdermal testosterone treatment in women with impaired sexual function after oophorectomy. N Engl J Med. 2000 Sep 7;343(10):682-8. doi: 10.1056/NEJM200009073431002. PMID 10974131
- [Background] Gleicher N, Weghofer A, Barad DH. The role of androgens in follicle maturation and ovulation induction: friend or foe of infertility treatment? Reprod Biol Endocrinol. 2011 Aug 17;9:116. doi: 10.1186/1477-7827-9-116. PMID 21849061
- [Background] Zhang HH, Xu PY, Wu J, Zou WW, Xu XM, Cao XY, Wei LZ. Dehydroepiandrosterone improves follicular fluid bone morphogenetic protein-15 and accumulated embryo score of infertility patients with diminished ovarian reserve undergoing in vitro fertilization: a randomized controlled trial. J Ovarian Res. 2014 Oct 21;7:93. doi: 10.1186/s13048-014-0093-3. PMID 25330837
- [Background] Gleicher N, Weghofer A, Barad DH. Defining ovarian reserve to better understand ovarian aging. Reprod Biol Endocrinol. 2011 Feb 7;9:23. doi: 10.1186/1477-7827-9-23. PMID 21299886
- [Background] Casson PR, Santoro N, Elkind-Hirsch K, Carson SA, Hornsby PJ, Abraham G, Buster JE. Postmenopausal dehydroepiandrosterone administration increases free insulin-like growth factor-I and decreases high-density lipoprotein: a six-month trial. Fertil Steril. 1998 Jul;70(1):107-10. doi: 10.1016/s0015-0282(98)00121-6. PMID 9660430
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Mutlu MF, Erdem M, Erdem A, Yildiz S, Mutlu I, Arisoy O, Oktem M. Antral follicle count determines poor ovarian response better than anti-Mullerian hormone but age is the only predictor for live birth in in vitro fertilization cycles. J Assist Reprod Genet. 2013 Jun;30(5):657-65. doi: 10.1007/s10815-013-9975-3. Epub 2013 Mar 19. PMID 23508679
- [Background] Gleicher N, Barad DH. Dehydroepiandrosterone (DHEA) supplementation in diminished ovarian reserve (DOR). Reprod Biol Endocrinol. 2011 May 17;9:67. doi: 10.1186/1477-7827-9-67. PMID 21586137
- [Background] Casson PR, Lindsay MS, Pisarska MD, Carson SA, Buster JE. Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series. Hum Reprod. 2000 Oct;15(10):2129-32. doi: 10.1093/humrep/15.10.2129. PMID 11006185
- [Background] Mamas L, Mamas E. Dehydroepiandrosterone supplementation in assisted reproduction: rationale and results. Curr Opin Obstet Gynecol. 2009 Aug;21(4):306-8. doi: 10.1097/gco.0b013e32832e0785. PMID 19610174
- [Background] Sunkara SK, Pundir J, Khalaf Y. Effect of androgen supplementation or modulation on ovarian stimulation outcome in poor responders: a meta-analysis. Reprod Biomed Online. 2011 Jun;22(6):545-55. doi: 10.1016/j.rbmo.2011.01.015. Epub 2011 Feb 17. PMID 21493151
- [Background] Gleicher N, Weghofer A, Barad DH. Dehydroepiandrosterone (DHEA) reduces embryo aneuploidy: direct evidence from preimplantation genetic screening (PGS). Reprod Biol Endocrinol. 2010 Nov 10;8:140. doi: 10.1186/1477-7827-8-140. PMID 21067609
- [Background] Ferrario M, Secomandi R, Cappato M, Galbignani E, Frigerio L, Arnoldi M, Fusi FM. Ovarian and adrenal androgens may be useful markers to predict oocyte competence and embryo development in older women. Gynecol Endocrinol. 2015 Feb;31(2):125-30. doi: 10.3109/09513590.2014.964639. Epub 2014 Sep 26. PMID 25259725
- [Background] Weissman A, Horowitz E, Ravhon A, Levran D. Administration of DHEA augments progesterone production in a woman with low ovarian reserve being transplanted with cryopreserved ovarian tissue. J Assist Reprod Genet. 2014 Nov;31(11):1565. doi: 10.1007/s10815-014-0358-1. Epub 2014 Oct 3. No abstract available. PMID 25278174
- [Background] Pediaditakis I, Iliopoulos I, Theologidis I, Delivanoglou N, Margioris AN, Charalampopoulos I, Gravanis A. Dehydroepiandrosterone: an ancestral ligand of neurotrophin receptors. Endocrinology. 2015 Jan;156(1):16-23. doi: 10.1210/en.2014-1596. PMID 25330101
- [Background] Cecconello AL, Trapp M, Hoefel AL, Marques CV, Arbo BD, Osterkamp G, Kucharski LC, Ribeiro MF. Sex-related differences in the effects of high-fat diets on DHEA-treated rats. Endocrine. 2015 Apr;48(3):985-94. doi: 10.1007/s12020-014-0396-6. Epub 2014 Oct 10. PMID 25300783
- [Background] Buster JE. Transvaginal dehydroepiandrosterone: an unconventional proposal to deliver a mysterious androgen that has no receptor or target tissue using a strategy with a new name: hormone precursor replacement therapy (HPRT). Menopause. 2009 Sep-Oct;16(5):858-9. doi: 10.1097/gme.0b013e3181ae1fca. No abstract available. PMID 19574935
- [Result] Artini PG, Simi G, Ruggiero M, Pinelli S, Di Berardino OM, Papini F, Papini S, Monteleone P, Cela V. DHEA supplementation improves follicular microenviroment in poor responder patients. Gynecol Endocrinol. 2012 Sep;28(9):669-73. doi: 10.3109/09513590.2012.705386. Epub 2012 Jul 26. PMID 22835219
- [Result] Barad D, Brill H, Gleicher N. Update on the use of dehydroepiandrosterone supplementation among women with diminished ovarian function. J Assist Reprod Genet. 2007 Dec;24(12):629-34. doi: 10.1007/s10815-007-9178-x. Epub 2007 Dec 11. PMID 18071895
- [Result] Gleicher N, Ryan E, Weghofer A, Blanco-Mejia S, Barad DH. Miscarriage rates after dehydroepiandrosterone (DHEA) supplementation in women with diminished ovarian reserve: a case control study. Reprod Biol Endocrinol. 2009 Oct 7;7:108. doi: 10.1186/1477-7827-7-108. PMID 19811650
- [Result] Gleicher N, Weghofer A, Barad DH. Improvement in diminished ovarian reserve after dehydroepiandrosterone supplementation. Reprod Biomed Online. 2010 Sep;21(3):360-5. doi: 10.1016/j.rbmo.2010.04.006. Epub 2010 Apr 18. PMID 20638339
- [Result] Wiser A, Gonen O, Ghetler Y, Shavit T, Berkovitz A, Shulman A. Addition of dehydroepiandrosterone (DHEA) for poor-responder patients before and during IVF treatment improves the pregnancy rate: a randomized prospective study. Hum Reprod. 2010 Oct;25(10):2496-500. doi: 10.1093/humrep/deq220. Epub 2010 Aug 21. PMID 20729538
- [Result] Yilmaz N, Uygur D, Inal H, Gorkem U, Cicek N, Mollamahmutoglu L. Dehydroepiandrosterone supplementation improves predictive markers for diminished ovarian reserve: serum AMH, inhibin B and antral follicle count. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(2):257-60. doi: 10.1016/j.ejogrb.2013.04.003. Epub 2013 May 9. PMID 23664458
- [Result] Singh N, Zangmo R, Kumar S, Roy KK, Sharma JB, Malhotra N, Vanamail P. A prospective study on role of dehydroepiandrosterone (DHEA) on improving the ovarian reserve markers in infertile patients with poor ovarian reserve. Gynecol Endocrinol. 2013 Nov;29(11):989-92. doi: 10.3109/09513590.2013.824957. Epub 2013 Sep 4. PMID 24004296
- [Result] Gleicher N, Kim A, Weghofer A, Shohat-Tal A, Lazzaroni E, Lee HJ, Barad DH. Starting and resulting testosterone levels after androgen supplementation determine at all ages in vitro fertilization (IVF) pregnancy rates in women with diminished ovarian reserve (DOR). J Assist Reprod Genet. 2013 Jan;30(1):49-62. doi: 10.1007/s10815-012-9890-z. Epub 2012 Dec 5. PMID 23212832
- [Result] Yeung TW, Li RH, Lee VC, Ho PC, Ng EH. A randomized double-blinded placebo-controlled trial on the effect of dehydroepiandrosterone for 16 weeks on ovarian response markers in women with primary ovarian insufficiency. J Clin Endocrinol Metab. 2013 Jan;98(1):380-8. doi: 10.1210/jc.2012-3071. Epub 2012 Nov 8. PMID 23144466
- [Result] Yeung TW, Chai J, Li RH, Lee VC, Ho PC, Ng EH. A randomized, controlled, pilot trial on the effect of dehydroepiandrosterone on ovarian response markers, ovarian response, and in vitro fertilization outcomes in poor responders. Fertil Steril. 2014 Jul;102(1):108-115.e1. doi: 10.1016/j.fertnstert.2014.03.044. Epub 2014 May 3. PMID 24796766
- [Result] Xu B, Li Z, Yue J, Jin L, Li Y, Ai J, Zhang H, Zhu G. Effect of dehydroepiandrosterone administration in patients with poor ovarian response according to the Bologna criteria. PLoS One. 2014 Jun 16;9(6):e99858. doi: 10.1371/journal.pone.0099858. eCollection 2014. PMID 24932478
- [Result] Barad D, Gleicher N. Effect of dehydroepiandrosterone on oocyte and embryo yields, embryo grade and cell number in IVF. Hum Reprod. 2006 Nov;21(11):2845-9. doi: 10.1093/humrep/del254. Epub 2006 Sep 22. PMID 16997936
- [Result] Jirge PR, Chougule SM, Gavali VG, Bhomkar DA. Impact of dehydroepiandrosterone on clinical outcome in poor responders: A pilot study in women undergoing in vitro fertilization, using bologna criteria. J Hum Reprod Sci. 2014 Jul;7(3):175-80. doi: 10.4103/0974-1208.142477. PMID 25395742